CLINICAL TRIAL: NCT06475586
Title: Effect of Semaglutide on the Inflammatory Response and Clinical Course of Psoriatic Lesions in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Semaglutide on the Psoriatic Lesions in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/4.48/23
Record Dates: First submitted 2024-06-11; First posted 2024-06-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis Vulgaris; Diabetes Type 2
Keywords: psoriasis; diabetes type 2; semaglutide; cytokine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Psoriasis | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double (participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- semaglutide (Experimental): The initial dose of the medicine is 0.25 mg once a week, for the duration of 4 weeks. Then the dose is increased to 0.5 mg per week, for the duration of 4 weeks. After at least 4 weeks, the dose can be increased from 0.5 mg to 1 mg per 4 week. Totally 12 weeks
  Interventions: Drug: Semaglutide
- controled group (No Intervention): Patients with DMT2 and psoriasis, who are already on metformin therapy in the maximally tolerated dose and other oral antidiabetics, except on therapy with GLP-1 RA and SGLT-2 inhibitors.

INTERVENTIONS:
Drug: Semaglutide — 0.25mg 4 weeks, 0.5mg per 4 weeks and 1.0mg per 4 weeks, totally 12 weeks
  Other Names: ozempic
  Arms: semaglutide

SUMMARY:
The use of semaglutide in patients with DMT2 and psoriasis contributes to improving the clinical picture of psoriasis and reducing the inflammatory response

DETAILED DESCRIPTION:
After being informed about the study and potential risiks all patients giving written informed consent will undergo a 1-week screening period to determine eliglibility for study entry at week 0, patients who meet the eligibility requirements will be randomized.

Study was conducted in two cohort Cohort 1. Patients with DMT2 and psoriasis, who are already on metformin therapy in the maximally tolerated dose and to whom semaglutide will be introduced into the therapy, in the maximum tolerated dose of semaglutide (0.25mg, 0.5mg per week or 1.0mg per week).

Cohort 2. Patients with DMT2 and psoriasis, who are already on metformin therapy in the maximally tolerated dose and other oral antidiabetics, except on therapy with GLP-1 RA and SGLT-2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed a personal consent to participate in the study,
* Patients with a typical clinical picture of moderately-severe to severe plaque psoriasis (PASI SCORE ≥10) and
* DMT2 diagnosed at least 6 months before inclusion in the study,
* Patients who were not treated with immunosuppressive therapy.

Exclusion Criteria:

* Other forms of psoriasis,
* Other chronic, inflammatory diseases (data obtained by reviewing the medical history),
* Drugs that can cause the appearance of psoriasis (lithium, systemic antimalarials, systemic corticosteroids) - for the past 3 months,
* Systemic therapy of vulgaris psoriasis 3 months before inclusion in the study,
* Patients on therapy with other GLP-1 RAs except semaglutide (liraglutide, dulaglutide, lixisenatide), SGLT-2 inhibitors (empagliflozin and dapagliflozin) and NSAIDs, photo UVB therapy,
* Patients who did not personally sign consent to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 30 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
clinical characteristics of patients with psoriasis | up to 12 weeks
  clinical examination by a dermatovenerologist (PASI SCORE- Psoriasis Area and Severity Index). To assess disease activity, i.e. skin surface affected by changes (erythema, infiltration and extent of squamous matter), investigators used the PASI score. According to the European consensus, mild psoriasis is defined as PASI≤10 and DLQI≤10, while moderate psoriasis is defined as PASi>10 and DLQI>10.
Determine BMI Body Mass Index | up to 12 weeks
  e.g., weight and height will be combined to report BMI in kg/m^2
Serum values of TNFa, IL-1b, IL-6, IL-17 and IL-23 | up to12 weeks
  ELISA-Enyzme linked immunosorbent assay technique -Bio Legend ELISA MAX Deluxe Sets, Bio Legend, San Diego, CA.
  same units
Correlation between the course and prognosis of the disease after the treatment | up to 12 weeks
  the Wilcoxon Mann-Whitney test for two independent groups will be used. Spearman's correlation analysis will be used to determine the correlation between parameters, binary logistic regression
Change in HgbA1C, | up to 12 weeks
  by enzymatic method with hexakinase glucose-6-phosphate dehydrogenase (Roche Diagnostic) will be expressed in %
lipid status, change in Total cholesterol (TC), low-density lipoprotein(LDL), high-density lipoprotein (HDL) and triglicerides | up to 12 weeks
  Biochemical analyses Clinical colorimetric tests, and results will be expressed in same units
fasting insulin | up to 12 weeks
  Biochemical analyses
Change in inflammation marker level: CRP, | up to 12 weeks
  Biochemical analyses-Turbid metric test
fasting glycemia | up to 12 weeks
  by enzymatic method with hexakinase glucose-6-phosphate dehydrogenase (Roche Diagnostic)
urate | up to 12 weeks
  Biochemical analyses

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Petkovic-Dabic, Principal Investigator — Faculty of Medicine Banja Luka
Locations (1):
- University of Banja Luka, Faculty of Medicine, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Result] Costanzo G, Curatolo S, Busa B, Belfiore A, Gullo D. Two birds one stone: semaglutide is highly effective against severe psoriasis in a type 2 diabetic patient. Endocrinol Diabetes Metab Case Rep. 2021 Aug 1;2021:21-0007. doi: 10.1530/EDM-21-0007. Online ahead of print. PMID 34463640
- [Result] Nauck MA, Quast DR, Wefers J, Meier JJ. GLP-1 receptor agonists in the treatment of type 2 diabetes - state-of-the-art. Mol Metab. 2021 Apr;46:101102. doi: 10.1016/j.molmet.2020.101102. Epub 2020 Oct 14. PMID 33068776

DOCUMENTS (3):
  • Study Protocol (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT06475586/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT06475586/SAP_001.pdf
  • Informed Consent Form (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT06475586/ICF_002.pdf